CLINICAL TRIAL: NCT04079114
Title: Post Market Clinical Follow-Up Study of the Zimmer Stafit Acetabular System. A Multicenter, Prospective, Non-controlled Study
Brief Title: Post Market Clinical Follow-Up of the Zimmer Stafit Acetabular System
Status: Terminated | Type: Observational
Why Stopped: Stafit Acetabular System not CE marked anymore
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 09H07
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Hip; Fracture of Hip; Avascular Necrosis of Hip; Dislocated Hip; Osteonecrosis; Post-traumatic; Arthrosis; Rheumatoid Arthritis; Subluxation Hip
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Fractures; Hip Dislocation; Osteonecrosis; Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Device: Patients who received the Stafit Acetabular System — Patients, suffering from severe hip pain and disability, requiring primary total hip arthroplasty with high risk of dislocation, who meet the inclusion/exclusion criteria.

SUMMARY:
This study is a Post Market Clinical Follow up study to fulfil the post market surveillance obligations according to Medical Device Directive and European Medical Device Vigilance System (MEDDEV) 2.12-2. The data collected from this study will serve the purpose of confirming safety and performance of the Zimmer Stafit Acetabular System.

DETAILED DESCRIPTION:
The objective of this study is to obtain implant survival and outcome data on the Stafit Acetabular System by analysis of standard scoring systems, radiographs, and adverse event records.

Data will be used to monitor pain, mobility, dislocation rate and implant survival, and to confirm the long-term safety and performance of the Stafit Acetabular System in primary total hip arthroplasty.

The study design is a multi-center, prospective, non-controlled, consecutive cohort post market clinical follow-up study, involving orthopedic surgeons skilled in total hip arthroplasty procedures and experienced with the Stafit Acetabular System.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Patients suffering from severe hip pain and disability requiring a primary total hip arthroplasty.
* 18 years minimum
* Patients able to participate in a follow-up program based upon physical examination and medical history
* Patients who have provided written informed consent by signing the Patient Informed Consent Form.

Exclusion Criteria:

* Patients who are unwilling or unable to give informed consent, or to comply with the follow-up program
* Known pregnancy
* Revision hip arthroplasty

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients, suffering from severe hip pain and disability, requiring primary total hip arthroplasty with high risk of dislocation, who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Study Director — Zimmer Biomet

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Who Received the Stafit Acetabular System
Started | 166
Completed | 0 (Study prematurely terminated.)
Not Completed | 166
Not completed — Study prematuely terminated. | 166

BASELINE CHARACTERISTICS:
Arm/Group | Patients Who Received the Stafit Acetabular System
Number analyzed (Participants) | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival
Description: Represents the implants that survived by counting the number of implants revised.
Time Frame: 3 years postoperatively, due to early study termination
Population: Outcome Measure Data at 3 years postoperative (Study early terminated). The Kaplan-Meier survival rate with cup revision for any reason.
Measure: Number; unit: percentage of implant survival
Units Other Than Participants: Implants
Arm/Group | Patients Who Received the Stafit Acetabular System
Number analyzed (Participants) | 80
Number analyzed (Implants) | 82
percentage of implant survival | 100

2. Primary Outcome: Dislocation Rate
Description: Assessed by counting the number of implant dislocations
Time Frame: 2 years
Population: Count of the number of dislocations 2 years postoperatively.
Measure: Number; unit: Implant Dislocations
Units Other Than Participants: implants
Arm/Group | Patients Who Received the Stafit Acetabular System
Number analyzed (Participants) | 161
Number analyzed (implants) | 166
Implant Dislocations | 0

3. Secondary Outcome: Evaluation of Pain and Functional Performance Determined by the Harris Hip Score
Description: The Harris Hip Score is a questionnaire filled by the surgeon on the patients who received a hip implant. The domains covered are pain, function, absence of deformity, and range of motion. The pain domain measures pain severity and its effect on activities and need for pain medication.
  The function domain consists of daily activities (stairs, public transportation, sitting, and managing shoes and socks) and gait (limp, support needed for walking, and walking distance). Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction.
  There are 10 items. The score has a minimum of 0 (worst possible score) to a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).
Time Frame: 3 years postoperatively, due to early study termination
Population: Outcome Measure Data at 3 years postoperative (Study early terminated). Number Of Unilateral Participants: 48 Unilaterals; Number Of Bilateral Participants : 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Patients Who Received the Stafit Acetabular System
Number analyzed (Participants) | 49
Number analyzed (Implants) | 50
score on a scale | 91.5 (10.3)

4. Secondary Outcome: Confirmation of Safety Based on Complications
Description: Reported number of patients with adverse events related to the implant. Adverse events include: dislocations of the hip, revisions and removals of the implants
Time Frame: 3 years postoperatively, due to early study termination
Population: Outcome Measure Data at 3 years postoperative (Study early terminated). Record of any adverse events related to the Stafit Acetabular System.
Measure: Number; unit: study patients
Arm/Group | Patients Who Received the Stafit Acetabular System
Number analyzed (Participants) | 166
study patients | 1

ADVERSE EVENTS:
Time Frame: follow-up visits at 6-12 weeks, 1, 2, and up to 3 years postoperatively.
Description: List of all the adverse events reported until the early study termination (some patients came until 3 year follow-up).
Arm/Group | Patients Who Received the Stafit Acetabular System
All-Cause Mortality (participants affected / at risk) | 6/166
Serious Adverse Events (participants affected / at risk) | 10/166
Other Adverse Events (participants affected / at risk) | 11/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Who Received the Stafit Acetabular System (N=166)
Femoral Implant Fracture (Surgical and medical procedures) | 1 — Treated by change of the Stem
Death (Stroke) (Blood and lymphatic system disorders) | 1
Death (General disorders) | 1
Infection (Infections and infestations) | 1 — Treated by lavage and antibiotic.
Deep Infection <6 Weeks (Infections and infestations) | 1 — Treated by lavage and antibiotic.
Infection (Infections and infestations) | 1 — Treated by 2 Red cell transfusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Who Received the Stafit Acetabular System (N=166)
Deep Infection <6 Weeks (Infections and infestations) | 1 — Treated by lavage and antibiotic
Stroke (Blood and lymphatic system disorders) | 1
Peroperative fracture of the femur (Surgical and medical procedures) | 1 — Treated by peroperative cerclage of the femur.
Vascular Injury (Vascular disorders) | 1 — Treated by suture and vascular surgical exploration
Fracture femur (Surgical and medical procedures) | 1 — Treated by plate osteosynthesis.
Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 1 — Treated by implantation of a nail.
Suspicion infection (Infections and infestations) | 1 — Hospitalization
Axonal mononeuropathy (Nervous system disorders) | 1 — Treated by move of the knee.
Total Knee Arthroplasty Left (Surgical and medical procedures) | 1
Fall (Social circumstances) | 1
Fracture of Trochanter (Surgical and medical procedures) | 1 — Treated by Cerclage
Haematoma (Blood and lymphatic system disorders) | 1 — Treated by Lavage and antibiotic
Cardiac Arrhythmia (Cardiac disorders) | 1 — Treated by change of the heart treatment.
Transfusion Reaction (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Early study termination leading less patients enrolled and shorter follow-up as initially planned in the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT04079114/Prot_SAP_000.pdf